CLINICAL TRIAL: NCT05893992
Title: Impacts of Hearing Aid Use on Listening Effort and Motivation Using fNIRS
Brief Title: fNIRS, Listening Effort, and Motivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: Toronto Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SRF-15557
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2023-05

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids; Auscultation

STUDY DESIGN:
Intervention Model Description: A single cohort of participants will receive and be assessed in all treatment/intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital noise management, then quiet listening (Experimental): Participants with hearing loss who are candidates for hearing aids first listen using the device for hearing loss compensation with digital noise management features, followed by the device for hearing loss compensation for listening in quiet environments.
  Interventions: Device: Hearing aids with noise management features for listening in noise; Device: Hearing aid for listening in quiet environments
- Quiet listening, then digital noise management (Experimental): Participants with hearing loss who are candidates for hearing aids first listen using the device for hearing loss compensation for listening in quiet environments, followed by the device for hearing loss compensation with digital noise management features.
  Interventions: Device: Hearing aids with noise management features for listening in noise; Device: Hearing aid for listening in quiet environments

INTERVENTIONS:
Device: Hearing aids with noise management features for listening in noise — Device for hearing loss compensation with digital noise management features
Device: Hearing aid for listening in quiet environments — Device for hearing loss compensation for listening in quiet environments

SUMMARY:
The purpose of the current study is to measure oxygenation in the PFC using fNIRS in a sample of older adults with hearing loss. Participants will be instructed to listen to sentences in noise at a challenging signal-to-noise-ratio, and to repeat the word that they heard and rate how much subjective listening effort was required in order to make out the words. fNIRS will be measured throughout. Participants will complete the task using a hearing aid program intended for listening in quiet, and a hearing aid program with new advanced noise management features.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-99) years
* Binaural, symmetrical, sensorineural N2 (mild) to N5 (moderate-severe) hearing loss
* Fluent in English

Exclusion Criteria:

* Minors (17 years or less)
* Not able to tolerate wearing of hearing aids
* Vulnerable populations

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-09-23 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jinyu Qian, PhD, Principal Investigator — Sonova AG
Locations (1):
- Sonova Innovation Centre Toronto, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Digital Noise Management, Then Quiet Listening | Quiet Listening, Then Digital Noise Management
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Hearing Loss: All participants will have hearing loss and be assigned to all two interventions. The interventions consist of calm-situation listening and noise management feature.
  Hearing aids with noise management features for listening in noise: Device for hearing loss compensation with digital noise management features
  Hearing aid for listening in quiet environments: Device for hearing loss compensation for listening in quiet environments
Arm/Group | Hearing Loss
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 26

OUTCOME MEASURES:

1. Primary Outcome: Oxygenation Using Functional Near Infrared Spectroscopy (fNIRS)
Description: Infrared light scattered from the prefrontal cortex, which is indicative of concentration of oxygenated blood in that region. fNIRS in the prefrontal cortex is intended to index both motivation and listening effort.
Time Frame: Session 1, 2, 3 and 4; assessed for up to 2 hours
Measure: Mean (Standard Error); unit: Oxygenation (uMol)
Groups:
- Participants With Hearing Loss: Participants with hearing loss who are candidates for hearing aids
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 26
Oxygenation (uMol)
  Hearing aid with noise management | -14.85 (4.65)
  Hearing aids for quiet listening | 4.15 (4.65)

2. Secondary Outcome: Listening Accuracy
Description: Speech understanding in noise percent correct scores
Time Frame: Session 1, 2, 3 and 4; assessed for up to 2 hours
Measure: Mean (Standard Deviation); unit: Percentage of words repeated correctly
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 26
Percentage of words repeated correctly
  Hearing aids with noise management | 75.8 (15.2)
  Hearing aids for quiet listening | 62.3 (19.4)

3. Secondary Outcome: Subjective Listening Effort Rating
Description: Participants rate how much listening effort was required in order to make out a sentence from 1-7, where lower scores mean less effort required.
Time Frame: Session 1, 2, 3 and 4; assessed for up to 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 26
units on a scale
  Hearing aids with noise management | 3.08 (0.960)
  Hearing aids for quiet listening | 4.08 (0.892)

ADVERSE EVENTS:
Time Frame: Session 1, 2, 3 and 4; assessed for up to 2 hours
Arm/Group | Hearing Loss
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT05893992/Prot_SAP_000.pdf